CLINICAL TRIAL: NCT04078321
Title: Evaluation of Multifocal Transcutaneous Electrical Stimulation for Self-treatment Among Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mollii
Record Dates: First submitted 2019-08-23; First posted 2019-09-06 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2021-01

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Single case studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single case design (Experimental): Single case studies
  Interventions: Other: Mollii ®

INTERVENTIONS:
Other: Mollii ® — The garment claims to have a 48 hours lasting effect of an hour of treatment. The garment should be worn for at least 1 hour every other day. All participants receive individually tailored garments and individually tailored appropriate training towards specific goals set in connection to study start. The garment is used in the home environment and the family is responsible for documentation of use in a diary. Measurements is performed following an ABAB design for four weeks. Measurement performed at 12 occasions during the four weeks are; spasticity, physical function, pain, sleep and adherence. Standardized protocols for the intervention are provided to involved physical therapists.

SUMMARY:
The main purpose with this study is to investigate the effectiveness of a garment with integrated electrodes for multifocal transcutaneous electrical stimulation intended for treatment of spasticity in children with cerebral palsy.

DETAILED DESCRIPTION:
The effect and use of the garment will be evaluated in single - case studies using ABAB design.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy diagnosis, with spasticity as the main symptom
* Established GMFCS, levels 1-5
* MACS level, levels 1-5
* Included in the CPUP * national quality register
* Person should be between 4 years and up to 18 years
* Secured communication to and from person
* Neing able to convey pain or discomfort.

Exclusion Criteria:

* No treatment received within next three months before participation with botulinum toxin treatment to reduce spasticity.
* The patient may not have a shunt or other medical pump that may be affected by the electrical stimulation provided by the garment.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | four weeks
  Measures of spasticity at 12 Occasions using the Modified Ashworth Scale. Measures include both upper and lower limbs. Scores are rated by::
  0= No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+= Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
  The mesures will be perfomed three times each week for four weeks.

SECONDARY OUTCOMES:
Timed Up and Go (time) | four weeks
  Measures of physical function at 12 Occasions, the mesures will be perfomed three times each week for four weeks.
  Instructions:
  The patient should sit on a standard armchair, placing his/her back against the chair and resting his/her arms chair's arms. Any assistive device used for walking should be nearby. Regular footwear and customary walking aids should be used. The patient should walk to a line that is 3 meters (9.8 feet) away, turn around at the line, walk back to the chair, and sit down. The test ends when the patient's buttocks touch the seat. Patients should be instructed to use a comfortable and safe walking speed. A stopwatch should be used to time the test (in seconds).
Faces pain scale 0-5 | four weeks
  Measures of pain recorded daily in a diary. Rating 0 indicating
Two questions of sleeling quality, three answer options provided | four weeks
  Measures of sleep recorded daily in a diary
Adherence measured by days using the garment during the intervention | four weeks
  The participant will report in a diary each day the garment is used and the diary also provide the possibility to add a comment.
Level of Sitting Scale (score 1-8) | four weeks
  Measures of physical function at 12 Occasions, the mesures will be perfomed three times each week for four weeks.
  The participant will be placed in sitting position. Score 1 indicating lowest score on sitting function (highest need of support) and 8 indicating highest function on sitting function (lowest need of support)
Box and block test (number of blocks moved in one minute) | four weeks
  Measures of physical function at 12 Occasions, the mesures will be perfomed three times each week for four weeks.The score is the number of blocks carried from one compartment to the other in one minute. Score each hand separately.
  After testing, the examiner should count the blocks If a patient transports two or more blocks at the same time, this should be noted and the number subtracted from the total.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Arkkukangas, PhD, Study Director — Research and Development in Sörmland
Locations (1):
- Marina Arkkukangas, Eskilstuna, Sweden

IPD SHARING:
Plan to Share IPD: No